CLINICAL TRIAL: NCT05945394
Title: The Surem TRAF3IP2 Level and Atherosclerotic Plaque Development in Human
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jin Geng, associate doctor, Nanjing Medical University
Other Study IDs: 20230503
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Heart Disease, Susceptibility to, 1
Keywords: TRAF3IP2, Coronary angiography, coronary deart disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The blood sample will be collected, and the surem TRAF3IP2 levels will be measured using ELASA.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected CHD who experienced CAG: Patients with suspected coronary heart disease who experienced coronary angiography
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an obvertional study, and there is no intervention.

SUMMARY:
To evaluate the association of surem TRAF3IP2 levels with the atherosclerotic plaque development in human

DETAILED DESCRIPTION:
Previous study had concluded that TRAF3IP2 plays a causal role in atherosclerotic plaque development and vulnerability in mice. However, no human data was available. In the present study, patients who receive coronary angiography will be enrolled. Their surem TRAF3IP2 levels will be tested using ELASA. The association of surem TRAF3IP2 levels with the atherosclerotic plaque will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected coronary heart disease
2. patients received coronary angiography

Exclusion Criteria:

1. NYHA III-IV
2. malignant tumor
3. acute infection
4. thyroid dysfunction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected coronary heart disease who experienced coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
stenosis of coronary artery | 1 week
  The stenosis of coronary artery based on the results of coronary angiography

SECONDARY OUTCOMES:
coronary artery calcium | 1 week
  The coronary artery calcification based on the results of coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Ma Shuren, MD, Study Director — NJMU
Locations (1):
- Huai'an First People's Hospital, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No